CLINICAL TRIAL: NCT06693505
Title: Cognitive Performance and Sleep Quality Following Caffeinated Chewing Gum in Night-shift Emergency Physicians: A Double-blind Randomized Crossover Controlled Trial
Brief Title: The Effect of Caffeinated Chewing Gum on Cognitive Performance in Night-shift Emergency Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, SHIH HAO WU, Clinical Assistant Professor, China Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Caffeinated Chewing Gum on EP
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Performance; Sleep Quality
Keywords: night shift worker; sleep deprivation; Reaction time; Stoop test; Visual search; Patient safety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: A Double-blind Randomized Crossover Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine trial (CAF) (Experimental): caffeinated chewing gum first, then followed with placebo gum, at least four weeks later Each trial was separated by at least four weeks to avoid interactive effects.
  Interventions: Combination Product: caffeinated chewing gum
- placebo trial (PL) (Placebo Comparator): placebo gum first, then followed with caffeinated chewing gum, at least 4 weeks later. Each trial was separated by at least four weeks to avoid interactive effects.
  Interventions: Combination Product: placebo

INTERVENTIONS:
Combination Product: caffeinated chewing gum — two pieces of caffeinated chewing gum at an absolute dose of 200 mg (Military Energy Gum®, Ford Gum and Machine Go, Akron, NY, USA)
  Arms: caffeine trial (CAF)
Combination Product: placebo — two pieces of similar looking and tasting placebo gum that did not contain caffeine (xylitol, lime mint, green; Lotte, Saitama, Japan) (PLA trial)
  Arms: placebo trial (PL)

SUMMARY:
This study aimed to examine the impact of caffeinated chewing gum on the cognitive performance of night-shift emergency physicians in a partially sleep-deprived state. A randomized, double-blind crossover controlled experimental design was employed in which fourteen (Age: 29.9 ± 1.44; height: 176.5±5.3; weight: 78.1±13.4) emergency physicians consumed either caffeinated chewing gum (CAF) containing 200 mg caffeine or a caffeine-free placebo gum (PLA) for 10 minutes at 03:30 am during their first 8-hour night shift after at least one day off, and completed cognitive performance tests before shift, mid-shift (10 minutes after gum chewing), and after shift, including included Corsi block test, Task-switching paradigm, Stroop Test, Visual search, and Wisconsin Card Sorting Task. Sleep quality was assessed subjectively by a single question score, and objectively by ActiGraph for one night on the off day and the last sleep before the first night shift, to evaluate the effect of sleep quality on cognitive performance.

DETAILED DESCRIPTION:
Methods 2.1. Design This experiment was a double-blind, repeated-measures, crossover design according to the guidelines of CONSORT 2010 and was divided into either a caffeine trial (CAF) or a placebo trial (PL). To eliminate the impact of individual physical differences, a crossover trial was conducted with the same group of subjects. Randomized groups were created using Microsoft 365-Excel (Microsoft, Redmond, Washington, United States), and allocation was randomized and unpredictable. Each trial was separated by at least four weeks to avoid interactive effects. This study compared CAF and PL trial to determine the effects of caffeinated chewing gum on cognitive performance in emergency physicians engaged in night shift work., and subjective, objective sleep quality. Caffeinated chewing gum and placebo chewing gum are very similar in appearance, color, size, shape, and flavor and are difficult to distinguish. The randomization was carried out by a research assistant, with another resident performing the experiment, and neither the subjects themselves nor the resident experimenting knew which group the subjects were assigned to or what type of gum they were assigned. Once the data has been collected, it will be forwarded to the group's statistical analyst for statistical analysis, who was also unaware of the group assignments. At least one week before the formal experiment, all subjects participated in three to five familiarization tests for the cognitive function tests. Sleep quality was also assessed subjectively by a single question score, and objectively by ActiGraph for one night on the off day and the last sleep before the first night shift. The primary outcome was the results of cognitive function tests, and the secondary outcome was the sleep quality.

2.2. Participants Fourteen healthy male emergency physicians were recruited in this study and based on previous research on caffeine in e-sport athletes, we used the G*power 3.1 software 24 to achieve an alpha value of 5% and a power of 0.8, which was sufficient for the study with only six subjects. However, due to the lack of relevant studies on the effects of caffeine and caffeinated chewing gum on cognitive functioning in night-shift healthcare workers, reference was made to a recent study that examined the cognitive performance of emergency physicians after 24 consecutive hours of on-call duty, which included 13 subjects. Therefore, it should be adequate to interpret the data derived and statistics from the study.

All participants had experience working regular rotating shifts on the emergency clinical front line and regularly accepted night shift assignments each month. The inclusion criteria were: (i) healthy male adults, those individuals who are free of pain, insomnia, or other injuries recently, without any medication used in recent 2 months, (ii) underwent rotating shifts on the emergency clinical front line with regularly accepted night shift more than two years. The exclusion criteria were: (i) allergy to caffeine, (ii) experience of adverse effects of caffeine, (iii) with cardiovascular diseases or any disease that made subjects feel ill. Two weeks before the main trial, all the participants were asked to avoid ingestion of more than 80 mg of caffeine a day. Before the experiment, all participants were fully informed of the experimental procedures and risks and provided informed consent. This study received approval from the Institutional Review Board of China Medical University Hospital (CMUH111-REC2-169). This study was conducted following the Declaration of Helsinki.

2.3. Protocol 2.3.1. Experimental procedure The entire study was conducted in the office of the emergency department of China Medical University Hospital, and the indoor ambient temperature was set at 22°C. Participants' diet and mealtimes were recorded for the 3 days before the first formal experiment, and the participants were required to follow the same diet 3 days before the next formal experiment. They were also required to avoid food and beverages with caffeine (e.g., coffee, energy drinks, chocolate, chocolate drink, and tea) 3 days before the formal experiment.

On the day of the formal experiment, participants had breakfast and lunch at 08:00 and 12:00, respectively. The participants arrived at the office at approximately 23:20 for the experiment. A brief explanation was given and the cognitive test was administered at 23:30, which took about 20 minutes to complete, after which the subjects were ready to go to work. At 03:30, according to the randomized results, the subjects were given two pieces of caffeinated chewing gum at an absolute dose of 200 mg (Military Energy Gum®, Ford Gum and Machine Go, Akron, NY, USA) (CAF trial) or two pieces of similar looking and tasting placebo gum that did not contain caffeine (xylitol, lime mint, green; Lotte, Saitama, Japan) (PLA trial). After 10 minutes of chewing, cognitive function tests were administered. Finally, the last cognitive function tests were performed after duty at 08:20. All subjects used a dedicated computer with a screen frame rate of at least 240 Hz and a mouse response rate of 1ms.

To explore the validity of the blinding method, we asked the participants (before and after the test) to identify the supplements they ingested. To do this, the question was as follows: "Which supplement do you think you ingested?" There are three possible answers to this question: (a) caffeine; (b) placebo; and (c) don't know. Furthermore, the occurrence of side effects or complications was recorded during the trial.

2.3.2. Outcome measure 2.3.2.1. Cognitive function tests Subjects were sequentially given five tests: Corsi block test, Task-switching paradigm, Stroop Test, Visual search, and Wisconsin Card Sorting Task. All the above cognitive function tests were conducted using Psych/Lab for Windows. Measures used in the literature have satisfactory reliability and validity.

2.3.2.1.1. Corsi block test There will be 9 purple squares in the screen, when the test starts, it will flash a number of them randomly in yellow color (the more the number increases), then you will hear "Go", then you have to click the order of the flashing ones, and then press "DONE" in the lower right corner. The smiley face means correct, the crying face means wrong. The maximum number of correct answers will be displayed at the end of the test, which is mainly to test the ability of situational awareness and working memory. The whole process takes about 2 minutes.

2.3.2.1.2. Task-switching paradigm There are two shapes (circle, square) and two colors (yellow, blue), four combinations in total. At the beginning of the test, you will see "SHAPE" or "COLOR" (which means that the answer to the question will be based on the shape or color), and then a colorful pattern (e.g., yellow square or blue circle) will appear, then answer the question according to the answer you have just seen (shape or color) as soon as possible. Press B for circles, N for squares, B for yellow, N for blue, and finally the average reaction speed is displayed, which is a test of cognitive structure, flexibility, and plasticity in task processing. The whole test takes about 4 minutes.

2.3.2.1.3. Stroop Test In this quiz, you will see different colors for different words, but all the answers are based on the colors (no matter what the words are). Press R for red, G for green, B for blue, and Y for yellow; for example, if you see "green in red color", you have to press R. The test results comprised a congruent condition, in which the key pressed corresponded correctly to the color on the screen, and an incongruent condition, in which the key pressed corresponded incorrectly to the color name on the screen. At the end of the test, the reaction time will be displayed, which is mainly a test of the ability to inhibit cognitive interference. The whole test takes about 5 minutes.

2.3.2.1.4. Visual search In the visual search test, participants identified orange "T" s on the screen from upside-down orange "T" s, blue "T" s, and upside-down blue "T" s. When an orange "T" would appear, the participants were required to press the spacebar as quickly as possible. If no orange "T" appeared, the participants were required to not react. The test contains 80 search displays, each containing 5, 10, 15 and 20 items, mainly to test the search ability of dynamic vision. Reaction speed was displayed at the end of the test, and the whole test took about 4 minutes.

2.3.2.1.5. Wisconsin Card Sorting Task There is a trial-and-error component to this test. You have to answer the questions first and then determine what the question is based on what is right or wrong. The test is presented in a matching mode, where a pattern on the left is matched with one of the four patterns on the right, and the matching criteria are color, shape, and number. During the test, the questions will be changed from time to time, so if you find out the rules and then suddenly get a question wrong, it means that the question has been changed. The number of errors is displayed at the end of the test to help measure a person's ability to reason abstractly and to change problem-solving strategies when necessary. The entire test lasted about 4 minutes.

2.3.2.2. Measure Of Sleep Participants wore a wrist ActiGraph (wActiSleep, Pensacola, Florida, United States) on the nondominant hand for 2 sleep periods, including the sleep on off day and the sleep before the first third night duty. The sleep data were obtained from ActiGraph monitors and analyzed by ActiLife software version 6 using the Cole-Kripke algorithm, including eight sleep indices (sleep latency, total counts, sleep efficiency, total sleep time [TST], wake after sleep onset [WASO], number of awakenings, length of awakenings, time in bed)[39, 40]. Participants also recorded the time they went to bed and woke up to enable coordinate checks with the actigraphic data. Daily sleep quality was measured using a question that was chosen because it was easy to conceptualize, simple to understand, and less burdensome for participants. The question asked was: On a scale of 0-10, with 0 being the worst sleep and 10 being the best, rate the quality of the previous sleep.

Participants self-reported age, marital status, exercise habits, smoking, caffeine and alcohol consumption, and chronic diseases. Height and weight were measured from which body mass index (BMI) was calculated as weight in kilograms divided by the square of height in meters (kg/m2).

Statistical analysis All data are presented as averages ± standard deviations. The Shapiro-Wilk test was used to examine the normality of the data. Cognitive performance, accuracy, and hit reaction time were analyzed through a paired sample t test. Effect sizes were calculated using Cohen's D. Tests were performed (t tests or χ2 tests) to test for differences at baseline between the two groups. A 2 × 2 mixed-design analysis of variance with repeated measures was used to examine the effects of the intervention. The Bang's Blinding Index (BBI ) was used to explore the effectiveness of the blinding whereas the McNemar test was used in the comparison of the incidence of side-effects between the placebo and caffeine conditions. All data were calculated using SPSS (version 20, Chicago, IL, USA), and the significance level was α < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* (i) healthy male adults, those individuals who are free of pain, insomnia, or other injuries recently, without any medication used in recent 2 months,
* (ii) underwent rotating shifts on the emergency clinical front line with regularly accepted night shift more than two years.

Exclusion Criteria:

* (i) allergy to caffeine,
* (ii) experience of adverse effects of caffeine,
* (iii) with cardiovascular diseases or any disease that made subjects feel ill.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Corsi block test | baseline (preintervention), immediately after the intervention
  There will be 9 purple squares in the screen, when the test starts, it will flash a number of them randomly in yellow color (the more the number increases), then you will hear "Go", then you have to click the order of the flashing ones, and then press "DONE" in the lower right corner. The smiley face means correct, the crying face means wrong. The maximum number of correct answers will be displayed at the end of the test, which is mainly to test the ability of situational awareness and working memory. The whole process takes about 2 minutes.
Task-switching paradigm | baseline (preintervention), immediately after the intervention
  There are two shapes (circle, square) and two colors (yellow, blue), four combinations in total. At the beginning of the test, you will see "SHAPE" or "COLOR" (which means that the answer to the question will be based on the shape or color), and then a colorful pattern (e.g., yellow square or blue circle) will appear, then answer the question according to the answer you have just seen (shape or color) as soon as possible. Press B for circles, N for squares, B for yellow, N for blue, and finally the average reaction speed is displayed, which is a test of cognitive structure, flexibility, and plasticity in task processing. The whole test takes about 4 minutes.
Stroop Test | baseline (preintervention), immediately after the intervention
  In this quiz, you will see different colors for different words, but all the answers are based on the colors (no matter what the words are). Press R for red, G for green, B for blue, and Y for yellow; for example, if you see "green in red color", you have to press R. The test results comprised a congruent condition, in which the key pressed corresponded correctly to the color on the screen, and an incongruent condition, in which the key pressed corresponded incorrectly to the color name on the screen. At the end of the test, the reaction time will be displayed, which is mainly a test of the ability to inhibit cognitive interference. The whole test takes about 5 minutes.
Visual search | baseline (preintervention), immediately after the intervention
  In the visual search test, participants identified orange "T" s on the screen from upside-down orange "T" s, blue "T" s, and upside-down blue "T" s. When an orange "T" would appear, the participants were required to press the spacebar as quickly as possible. If no orange "T" appeared, the participants were required to not react. The test contains 80 search displays, each containing 5, 10, 15 and 20 items, mainly to test the search ability of dynamic vision. Reaction speed was displayed at the end of the test, and the whole test took about 4 minutes.
Wisconsin Card Sorting Task | baseline (preintervention), immediately after the intervention
  There is a trial-and-error component to this test. You have to answer the questions first and then determine what the question is based on what is right or wrong. The test is presented in a matching mode, where a pattern on the left is matched with one of the four patterns on the right, and the matching criteria are color, shape, and number. During the test, the questions will be changed from time to time, so if you find out the rules and then suddenly get a question wrong, it means that the question has been changed. The number of errors is displayed at the end of the test to help measure a person's ability to reason abstractly and to change problem-solving strategies when necessary. The entire test lasted about 4 minutes.

SECONDARY OUTCOMES:
subjectively sleep quality | baseline (the sleep before intervention),the sleep after the intervention
  subjectively by a single question score
objectively sleep quality | baseline (the sleep before intervention),the sleep after the intervention
  objectively by ActiGraph

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
provide email on published journal, researcher who are interested , could mail to corresponding author and request the data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after published , for 5 years
Access Criteria: provide email on published journal, researcher who are interested , could mail to corresponding author and request the data

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT06693505/Prot_SAP_000.pdf